CLINICAL TRIAL: NCT05120323
Title: Video Directly Observed Therapy (vDOT) to Improve Inhaler Technique Among Pediatric Patients With Newly Diagnosed Asthma
Brief Title: vDOT for Newly Diagnosed Pediatric Asthma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Tamara Perry, Professor of Pediatrics, Chief, Allergy and Immunology Division, Arkansas Children's Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 273496
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Asthma in Children

STUDY DESIGN:
Intervention Model Description: They will be randomized to the intervention arm or standard of care arm.
Who Masked: Outcomes Assessor
Masking Description: The participants will have a follow up appointment at 3 months and the respiratory therapists will be blinded to the study treatment to assess the participant's inhaler technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vDOT Intervention Group (Experimental): The VDot group will submit videos via app to Emocha to have their inhaler technique graded to assess their inhaler technique.
  Interventions: Behavioral: vDOT Intervention Group
- Standard Asthma Care Group (No Intervention): Participants in the standard asthma care group will receive standard of care asthma education conducted by a respiratory therapist in the specialty clinics at Arkansas Children's Hospital at the baseline visit. Education will include standard of care instruction on the participant's prescribed asthma medications, how to use an asthma action plan, as well as training and demonstration of proper inhaler technique. They will not have any additional study activities until the 3-month visit. They will be instructed to take their medications as prescribed.

INTERVENTIONS:
Behavioral: vDOT Intervention Group — The vDOT intervention group will submit video clips of doses of inhaled controller asthma medication via the Emocha® smartphone application with each prescribed dose of inhaled controller medication. Each video will include a date and time stamp of the medication dose. Participant videos will be evaluated by trained personnel using an inhaler technique checklist to score each dose and create a report detailing the steps that were taken to complete the medication dose.
  Arms: vDOT Intervention Group

SUMMARY:
The goal of this research study is to compare the impact of video directly observed therapy on inhaler technique accuracy with participants receiving video directly observed therapy vs. participants receiving standard asthma care. Participants will be randomized between the two groups. We will follow up and compare the two groups to see if they have improved asthma control as measured by symptom-free days (SFD), higher inhaler technique at 3-month follow up, higher checklist scores on a standardized inhaler technique checklist, higher proportion of days covered (PDC) of their inhaled asthma controller medication, and have fewer acute care visits for asthma.

DETAILED DESCRIPTION:
Emocha® was originally developed by researchers at the Johns Hopkins University School of Medicine, the HIPAA-compliant platform was commercialized in 2014. Emocha® platform uses virtual communication tools (e.g. asynchronous video technology and secure 2-way messaging) to support and encourage adherence through timely feedback and positive reinforcement: helping users develop healthy behaviors and maintain high levels of medication adherence. The company leverages a public health practice called Directly Observed Therapy (DOT). DOT is a Center for Disease Control (CDC)-endorsed model of care that has been used by public health departments for decades to contain deadly infectious diseases.

Our overarching hypothesis is that compared to standard asthma medication education, vDOT will improve accuracy of inhaler technique (primary aim) and improve clinical outcomes such as medication adherence and asthma symptoms among children newly referred to asthma specialty clinic or those with a new inhaled asthma medication inhaler type.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 6 and ≤ 11 years old
2. Physician diagnosed persistent asthma (any severity) and verified by review of electronic medical record
3. New patient with a new prescription for inhaled preventive asthma medication referred to an asthma subspecialty clinic at Arkansas Children's OR established patient in the asthma, allergy or pulmonary subspecialty clinic with a new prescription for inhaled preventive asthma medication.
4. Regular access to Wi-Fi

Exclusion Criteria:

1. Significant underlying respiratory disease other than asthma such as cystic fibrosis
2. Significant co-morbid conditions, such as moderate to severe developmental delay that could interfere with the ability to communicate via interactive video
3. Current smoker
4. Caregiver/patient does not have access to a smartphone compatible with the Emocha® smartphone application
5. Caregiver and patient speaks and understands English as their primary language.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Inhaler technique | 3 months
  For all participants, the inhaler technique checklist will be completed at the baseline and 3-month visits. The rate of inhaler technique accuracy (absence of errors, yes/no) at 3-months will be compared between the vDOT intervention and standard asthma care groups (primary outcome). The number and type of technique errors for both groups will be recorded at 3-months. b. For intervention participants only, each (daily) submitted video will receive 2 ratings to record a numeric score (0-10) and a yes/no accuracy score. The number and type of technique errors (i.e. did not shake inhaler, did not hold breath, etc) during the first 30 days will be assessed. The length of time to technique mastery (technique accuracy doses x 3 consecutive doses) will be recorded.
Symptom-free days | 3 months
  We will measure the change from baseline in the number of SFD during the prior 2 weeks, assessed at the end of the 3-month intervention period. This outcome measure is consistent with the symptom monitoring suggested by the national guidelines for asthma care and has been suggested as an appropriate surrogate marker for asthma control. We will ask parents to report the number of days during the prior 2 weeks that their child experienced no symptoms of asthma (defined as a 24 hour period with no coughing, wheezing, chest tightness, or shortness of breath, and no need for rescue medications).
Healthcare utilization | 3 months
  Questions regarding healthcare utilization and asthma exacerbations will be included. We will ask caregivers to report the number of steroid bursts, unscheduled (acute) healthcare visits, emergency room visits, and hospitalizations due to asthma in the past 3 months at the baseline and 3-month visit.
Medication Adherence | 3 months
  As a proxy of medication adherence, we will measure the proportion of days covered (PDC) of their inhaled asthma medication for the 90 days (3 months) while enrolled in the proposed study.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara T. Perry, MD, Principal Investigator — University of Arkansas for Medical Sciences and Arkansas Children's Research Institute
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers. Only study staff will have access to individual participant data.